CLINICAL TRIAL: NCT00532675
Title: A Phase Ib, Multi-center, Open-label, Dose-escalation Study of Oral LBH589 When Administered in Combination With Oral Lenalidomide & Dexamethasone in Adult Patients With Multiple Myeloma
Brief Title: Safety Study of LBH589 When Given in Combination With Lenalidomide and Dexamethasone in Adult Patients With Multiple Myeloma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2206; 2006-007030-35 (EudraCT Number)
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Lenalidomide; Revlimid; Dexamethasone; LBH589; Combination
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Panobinostat; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PAN 5 mg (Experimental): Panobinostat 5 mg
  Interventions: Drug: LBH589; Combination Product: Lenalidomide
- PAN 10 mg (Experimental): Panobinostat 10 mg
  Interventions: Drug: LBH589; Combination Product: Lenalidomide
- PAN 20 mg (Experimental): Panobinostat 20 mg
  Interventions: Drug: LBH589; Combination Product: Lenalidomide
- PAN 25 mg (Experimental): Panobinostat 25 mg
  Interventions: Drug: LBH589; Combination Product: Lenalidomide

INTERVENTIONS:
Drug: LBH589 — PAN 5 mg and PAN 20 mg capsules
  Other Names: Panobinostat, PAN
Combination Product: Lenalidomide — Lenalidomide 5mg or 25 mg

SUMMARY:
This study will evaluate the safety of LBH589 given in combination with lenalidomide and dexamethasone in adult patients with multiple myeloma

ELIGIBILITY:
Inclusion criteria:

* Patients must have a diagnosis of active multiple myeloma
* Patients must have received at least one prior line of therapy and their disease has relapsed..
* Patients must be suitable for treatment with lenalidomide & dexamethasone.
* Adults ≥ 18 years old
* ECOG Performance Status ≤ 2
* Life expectancy > 12 weeks
* Patients must have acceptable neutrophil and platelet counts as well as adequate kidney and liver function.
* Able to sign informed consent and to comply with the protocol

Exclusion criteria:

* Primary refractory MM
* Peripheral neuropathy ≥ CTCAE grade 2
* Impaired cardiac function or clinically significant cardiac diseases
* Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
* Patients with diarrhea > CTCAE grade 1
* Patients using medications that have a relative risk of prolonging the QT interval
* Concomitant use of CYP3A4 inhibitors
* Patients with a history of deep vein thrombosis or thromboembolism within < 6 months prior to starting study treatment
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using 2 reliable forms of birth control
* Male patients whose sexual partners are WOCBP and who are unable to use a latex condom during sexual contact (even if they have undergone a vasectomy)
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-04-22 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
To determine the highest and safest dose of LBH589 when it is administered in combination with lenalidomide & dexamethasone | 24 weeks

SECONDARY OUTCOMES:
Safety and tolerability assessed by monitoring of adverse events, serious adverse events and laboratory parameters To characterize the pharmacokinetic profile of the study treatment To characterize the pharmacodynamic profile of the study treatment | Da1 to Day 3 (week 1 of first cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - UCSF Medical Center, San Francisco, California
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Winship Cancer Inst., Atlanta, Georgia
  - St. Vincent's Comprehensive Cancer Center, New York, New York
- Australia (2):
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Prahran, Victoria
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Results for CLBH589B2206 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17260